CLINICAL TRIAL: NCT06760676
Title: A Multiple Tumor Species, Open and Multi-center Clinical Study of Alpaloritovorelli Antibodies (QL-1706) Combined with Pulsed Low Dose Rate External Irradiation (PLDR) for Disease Progression After Previous Anti-tumor Therapy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhou peijie 2024-ky-02
Record Dates: First submitted 2024-12-18; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer; Non Small Cell Lung Cancer; Cervical Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pulsed low dose rate radiotherapy (PLDR) combined with Alpaloritovorelli antibodies (QL-1706)) (Experimental)
  Interventions: Radiation: Pulsed low dose rate radiotherapy (PLDR); Drug: Alpaloritovorelli antibodies

INTERVENTIONS:
Radiation: Pulsed low dose rate radiotherapy (PLDR) — Radiation 5 times per week, 2Gy each time which divided into 10 pulse doses, each pulse interval was 3 minutes, the dose rate was 0.067 Gy/min, and each treatment time was 30 minutes.
Drug: Alpaloritovorelli antibodies — PLDR external irradiation therapy was administered simultaneously with 5mg/kg Alpaloritovorelli antibodies for a 3-week regimen, the following maintenance treatment was 2 years.

SUMMARY:
For the recurrent and metastatic tumors after first-line treatment (such as lung cancer, esophageal cancer and cervical cancer), the risk of conventional fractionated secondary radiotherapy is high because the tumor is close to the hollow organs (such as heart, lung and small intestine). According to previous studies, combined chemotherapy regimens are often used, but the disease control rate (DCR) is limited, and drug resistance and poor tolerance of patients are prone to occur. The immune checkpoint inhibitors (ICB) has been considered as a new strategy for maintenance treatment of patients with recurrent and metastatic tumors, but only some patients can respond for a long time. Therefore, how to improve the clinical response rate of ICB has become an urgent problem to be solved. Pulsed low dose rate radiotherapy (PLDR), a new radiotherapy technology emerging in recent years, is expected to become a new way to solve the above difficulties. Alpaloritovorelli antibodies (QL-1706) is a new type of combination antibody independently developed by Qilu Pharmaceutical Co., Ltd. It is composed of IgG4 antibody targeting PD-1 (ipalorimab), and IgG1 antibody targeting CTLA-4 (tuvonralimab) in a fixed proportion. It has the synergistic mechanism of blocking PD-1 and CTLA-4 at the same time. The combination of these two antibodies forms a powerful synergistic effect and forms positive feedback in the tumor immune cycle.

Pulsed low dose rate radiotherapy (PLDR) is a safe and feasible option for recurrent tumors with high risk of re-radiotherapy. It also has therapeutic advantages for refractory and massive tumors. The advantages of combined vascular targeting and chemotherapy have been initially demonstrated. As a new anti-tumor therapy, immunotherapy has shown clinical benefits in many types of cancer, but the overall effective rate is still limited, which may be due to the immune "desertification" of the tumor microenvironment. PLDR irradiation is expected to reverse the tumor inhibitory microenvironment by inducing the release of tumor associated antigen and increasing the killing function of T cells, activate tumor immunity and improve the response rate of immunotherapy. Based on this, this study plans to take the lead in carrying out this prospective clinical study through the combination of PLDR external irradiation and ICB treatment (QL-1706).

DETAILED DESCRIPTION:
For the recurrent and metastatic tumors after first-line treatment (such as lung cancer, esophageal cancer and cervical cancer), the risk of conventional fractionated secondary radiotherapy is high because the tumor is close to the hollow organs (such as heart, lung and small intestine). According to previous studies, combined chemotherapy regimens are often used, but the disease control rate (DCR) is limited, and drug resistance and poor tolerance of patients are prone to occur. The immune checkpoint inhibitors (ICB) has been considered as a new strategy for maintenance treatment of patients with recurrent and metastatic tumors, but only some patients can respond for a long time. Therefore, how to improve the clinical response rate of ICB has become an urgent problem to be solved. Pulsed low dose rate radiotherapy (PLDR), a new radiotherapy technology emerging in recent years, is expected to become a new way to solve the above difficulties. PLDR technology was first proposed by Tom é et al in 2007, and was first applied to the re-radiotherapy of recurrent tumors by Richards and Charlie Ma et al. The primary principle is the low-dose high radiosensitivity (HRS) of radiobiology, that is, a certain low-dose level of radiotherapy can increase the radiosensitivity of tumor cells and reduce the toxicity of normal tissues at the same time.

Alpaloritovorelli antibodies (QL-1706) is a new type of combination antibody independently developed by Qilu Pharmaceutical Co., Ltd. It is composed of IgG4 antibody targeting PD-1 (ipalorimab), and IgG1 antibody targeting CTLA-4 (tuvonralimab) in a fixed proportion. It has the synergistic mechanism of blocking PD-1 and CTLA-4 at the same time. The combination of these two antibodies forms a powerful synergistic effect and forms positive feedback in the tumor immune cycle. The combination antibody can maintain normal PD-1 antibody exposure in vivo and reduce the half-life of CTLA-4 antibody with lower toxicity and better tolerance. At present, sufficient preclinical studies of alpaloritovorelli antibodies have been completed, and a number of clinical studies are under way. The mechanism of action, safe dose range, mode of administration, toxicity characteristics and pharmacological characteristics are clear. Clinical research data show that the combination antibody of alpaloritovorelli is safe, controllable and tolerable in patients with solid tumors, and has shown encouraging efficacy in cervical cancer and other multiple tumors. Based on the results of DUBHE-C-206 trial, the combination antibody was approved by the China food and Drug Administration on September 30 of 2024, and the phase I safety test has been completed in the United States.

Pulsed low dose rate radiotherapy (PLDR) is a safe and feasible option for recurrent tumors with high risk of re-radiotherapy. It also has therapeutic advantages for refractory and massive tumors. The advantages of combined vascular targeting and chemotherapy have been initially demonstrated. As a new anti-tumor therapy, immunotherapy has shown clinical benefits in many types of cancer, but the overall effective rate is still limited, which may be due to the immune "desertification" of the tumor microenvironment. PLDR irradiation is expected to reverse the tumor inhibitory microenvironment by inducing the release of tumor associated antigen and increasing the killing function of T cells, activate tumor immunity and improve the response rate of immunotherapy. Based on this, this study plans to take the lead in carrying out this prospective clinical study through the combination of PLDR external irradiation and ICB treatment (QL-1706).

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined this study, signed informed consent, had good compliance, and were willing to cooperate with follow-up;
2. Male or female, age range of 18-75 years old (including 18 and 75 years old), gender not limited;
3. Confirmed by pathology as esophageal cancer, non-small cell lung cancer, or cervical cancer;
4. Expected survival period>3 months;
5. Patients who have progressed with first-line treatment in the past, (patients with local recurrence or distant metastasis of the tumor during (new) adjuvant therapy or ≤ 3 months after treatment are considered as first-line treatment)
6. ECOG score 0-2 points;
7. According to RECIST 1.1 criteria, there must be at least one measurable extracranial lesion;
8. The laboratory test results within one week before enrollment meet the following conditions: 1) Blood routine: HGB≥90g/L； WBC≥4.0×109/L； NEUT≥2.0×109/L； PLT ≥100×109/L； 2) Blood biochemistry: TBIL ≤ 1.5 × ULN; ALT and AST ≤ 3 × ULN (ALT and AST ≤ 5 × ULN in patients with liver metastases); BUN and Cr ≤ 1.5 × ULN and creatinine clearance rate ≥ 50 mL/min; 3) The results of cardiac ultrasound examination within the first two weeks of enrollment are consistent: left ventricular ejection fraction (LVEF)>50%;
9. Normal coagulation function, no active bleeding or thrombotic diseases;
10. Patients without contraindications for radiotherapy;
11. Patients of childbearing age who test negative for pregnancy and voluntarily adopt effective and reliable contraceptive measures during the trial period;
12. Subjects who have received anti-tumor treatment in the past should be enrolled only after the toxic reactions of previous treatment have stabilized and returned to baseline levels (except for residual hair loss effects) or after the CTCAE v5.0 rating score is ≤ 1.

Exclusion Criteria:

1. Patients with malignant tumors other than cervical cancer, esophageal cancer, and lung cancer;
2. In the first 5 years of randomization, patients with other active malignant tumors, except for locally curable tumors that have been cured, such as skin squamous cell carcinoma, skin basal cell carcinoma, superficial bladder cancer, and breast cancer in situ;
3. Patients who have participated in clinical trials of other drugs within the 4 weeks prior to enrollment, received radiation therapy targeting the target area within the 4 weeks prior to enrollment in this study, and received attenuated live vaccines within the 4 weeks prior to their first dose or planned to receive them during the study period; Within 4 weeks before the first administration, he received systematic treatment with traditional Chinese patent medicines and simple preparations with anti-tumor indications or Chinese herbal medicine with anti-tumor effect and drugs with immune regulation effect (such as thymosin, interferon, interleukin, etc.);
4. Within 6 months, there have been incidents of arterial/venous thrombosis, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
5. Simultaneously receiving any other anti-tumor treatment;
6. Individuals with a known history of allergies to the components of this medication regimen, a history of telangiectatic ataxia or other radiation hypersensitivity reactions;
7. Subjects with active infectious diseases;
8. Subjects with any severe and/or uncontrolled illnesses;
9. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results;
10. According to the investigator's judgment, there are concomitant diseases (including but not limited to severe hypertension, severe pulmonary dysfunction/disease, and severe diabetes beyond the control of drugs) that seriously endanger the patient's safety or affect the patient's completion of the study;
11. Having a clear history of neurological or mental disorders, including epilepsy or dementia, and being unable to cooperate with radiotherapy procedures;
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
13. Known history of interstitial lung disease or non infectious pneumonia;
14. Diagnosed with immunodeficiency or undergoing systemic corticosteroid therapy or any other form of immunosuppressive therapy, with active or potentially recurrent autoimmune diseases, except for vitiligo, hair loss, psoriasis, or eczema that do not require systemic treatment; Hypothyroidism caused by autoimmune thyroiditis only requires stable doses of hormone replacement therapy; Type I diabetes requiring only a stable dose of insulin replacement therapy.;
15. Suffering from active or documented inflammatory bowel disease (such as Crohn's disease, ulcerative colitis), and active diverticulitis. Clinical manifestations of gastrointestinal obstruction, or the need for routine parenteral fluid replacement, parenteral nutrition, or indwelling gastric tube;
16. There are symptomatic central nervous system (CNS) metastases, leptomeningeal metastases, or spinal cord compression caused by metastases prior to signing informed consent. Individuals without clinical symptoms, who have clinical and/or imaging evidence of stable condition, have stopped corticosteroid and anticonvulsant drug treatment for at least 2 weeks, and do not require further treatment (radiotherapy, surgical resection, and/or corticosteroid treatment) may participate in this study;
17. There are currently cases of third interstitial fluid accumulation that require local treatment such as repeated puncture and drainage due to poor clinical control;
18. Exclude subjects with any of the following cardiovascular diseases:

    1. Occurrence of myocardial infarction, unstable angina, pulmonary embolism, acute/persistent myocardial ischemia, cerebrovascular accident, transient ischemic attack, or other clinically significant/drug-induced arterial or venous thrombosis, embolism, or ischemic events within 6 months prior to the first administration;
    2. Past and/or current presence of NYHA class III-IV congestive heart failure;
    3. Previous and/or current severe arrhythmias requiring medication treatment;
    4. Before the first administration, the 12 lead ECG showed a mean QT interval (QTcF) of>470 ms.
19. The researchers believe that the patient is not suitable to participate in any other circumstances of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6-12 months
  The proportion of patients whose tumor volume shrinks by 30% and can be maintained for more than four weeks, which is the sum of complete remission and partial remission (CR+PR).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol